CLINICAL TRIAL: NCT03779334
Title: An Open-Label Study of Risdiplam in Infants With Genetically Diagnosed and Presymptomatic Spinal Muscular Atrophy
Brief Title: A Study of Risdiplam in Infants With Genetically Diagnosed and Presymptomatic Spinal Muscular Atrophy
Acronym: Rainbowfish
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN40703; 2018-002087-12 (EudraCT Number); 2023-506009-20-00 (EU CTIS Number)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Intervention Model Description: Open-label, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Risdiplam (Experimental): Participants will be enrolled to receive risdiplam orally once daily at a dose selected to achieve the targeted exposure range.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Risdiplam will be administered orally.
  Other Names: Evrysdi

SUMMARY:
A global study of oral risdiplam in pre-symptomatic participants with spinal muscular atrophy (SMA).

DETAILED DESCRIPTION:
The study is an open-label, single-arm, multicenter clinical study to investigate the efficacy, safety, pharmacokinetics, and pharmacodynamics of risdiplam in infants aged from birth to 6 weeks who have been genetically diagnosed with SMA but are not yet presenting with symptoms. There will be a screening, treatment, open-label extension (OLE) and a follow-up. All participants will receive risdiplam orally once daily for 2 years followed by an OLE phase of at least 3 years and a follow-up (if applicable), for a total treatment duration of at least 5 years for each participant enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged from birth (1 day) to 6 weeks (42 days) of age at the time of first dose (Day 1); a minimum age of 7 days at first dose is required for the first infant to be enrolled
* Gestational age of 37-42 weeks for singleton births; gestational age of 34-42 weeks for twins
* Body weight >= 3rd percentile for age, using appropriate country-specific guidelines
* Genetic diagnosis of 5q-autosomal recessive SMA, including confirmation of homozygous deletion or compound heterozygosity predictive of loss of function of the SMN1 gene
* Absence of clinical signs or symptoms at screening (Day -42 to Day -2) or at baseline (Day -1) that are, in the opinion of the investigator, strongly suggestive of SMA
* Receiving adequate nutrition and hydration at the time of screening, in the opinion of the investigator
* Adequately recovered from any acute illness at baseline and considered well enough to participate in the study, in the opinion of the investigator
* Able and expected to be able to safely travel to the study site for the entire duration of the study and in accordance to the frequency of required study visits, in the opinion of the investigator
* Able to complete all study procedures, measurements, and visits, and the parent (or caregiver), in the opinion of the investigator, has adequately supportive psychosocial circumstances
* Parent (or caregiver) is willing to consider nasogastric, naso-jejunal, or gastrostomy tube placement during the study to maintain safe hydration, nutrition, and treatment delivery, if recommended by the investigator
* Parent (or caregiver) is willing to consider the use of non-invasive ventilation during the study, if recommended by the investigator

Exclusion Criteria:

* Concomitant or previous participation in any investigational drug or device study at any time
* Concomitant or previous administration of an SMN2-targeting antisense oligonucleotide, SMN2-splicing modifier, or gene therapy either in a clinical study or as part of medical care
* Presence of significant concurrent syndromes or diseases
* In the opinion of the investigator, inadequate venous or capillary blood access for the study procedures
* Requiring invasive ventilation, tracheostomy or awake non-invasive ventilation
* Awake hypoxemia (SaO2 < 95%) with or without ventilator support
* Multiple or fixed contractures and/or hip subluxation or dislocation at birth
* Systolic blood pressure or diastolic blood pressure or heart rate considered to be clinically significant by the investigator
* Presence of clinically relevant ECG abnormalities before study drug administration; corrected QT interval using Bazett's method > 460 ms; personal or family history (first degree relatives) of congenital long QT syndrome indicating a safety risk for patients as determined by the investigator. First-degree atrioventricular block or isolated right bundle branch block are allowed
* The infant (and the mother, if breastfeeding the infant) taking any inhibitor of CYP3A4 taken within 2 weeks, any inducer of CYP3A4 taken within 4 weeks, any OCT 2 and MATE substrates within 2 weeks and known FMO1 or FMO3 inhibitors or substrates
* Clinically significant abnormalities in laboratory test results
* Ascertained or presumptive hypersensitivity to risdiplam or to the constituents of its formulation
* Treatment with oral salbutamol or another beta-2 adrenergic agonist taken orally for SMA is not allowed. Use of inhaled beta-2 adrenergic agonists is allowed
* Infants exposed to drugs with known retinal toxicity given to mothers during pregnancy (and lactation) should not be enrolled. Anticipated need for drugs known to cause retinal toxicity during the study.
* Diagnosis of ophthalmic diseases

Ages: 1 Day to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2027-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Nemours Children's Hospital, Orlando, Florida, United States
- Sydney Children's Hospital, Randwick, New South Wales, Australia
- Chr de La Citadelle, Liège, Belgium
- Hospital das Clinicas - FMUSP_X, São Paulo, São Paulo, Brazil
- Szpital Gdanskiego Uniwersytetu Medycznego, Gda?sk, Poland
- Russian Children Neuromuscular Center of Veltischev, Moscow, Moscow Oblast, Russia
- Kaohsiung Medical University Chung-Ho Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Finkel RS, Servais L, Vlodavets D, Zanoteli E, Mazurkiewicz-Beldzinska M, Jong YJ, Navas-Nazario A, Al-Muhaizea M, Araujo APQC, Nelson L, Wang Y, Jaber B, Gorni K, Kletzl H, Palfreeman L, Rabbia M, Summers D, Gaki E, Wagner KR, Fontoura P, Farrar MA, Bertini E; RAINBOWFISH Study Group. Risdiplam in Presymptomatic Spinal Muscular Atrophy. N Engl J Med. 2025 Aug 14;393(7):671-682. doi: 10.1056/NEJMoa2410120. PMID 40802943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 26 infants with spinal muscular atrophy (SMA) were enrolled in the study across 7 different sites in 7 countries.
Pre-assignment Details: The study enrolled infants aged from birth to 6 weeks who were genetically diagnosed with SMA but were not yet presenting with symptoms. Study arms were based on the number of copies of the SMN2 gene.
Groups:
- 2 SMN2 Copies, Risdiplam: Infants with 2 copies of SMN2 were enrolled to receive risdiplam orally once daily at a dose selected to achieve the targeted exposure range of close to 2000 ng*hr/mL.
- 3 SMN2 Copies, Risdiplam: Infants with 3 copies of SMN2 were enrolled to receive risdiplam orally once daily at a dose selected to achieve the targeted exposure range of close to 2000 ng*hr/mL.
- >/=4 SMN2 Copies, Risdiplam: Infants with 4 or more copies of SMN2 were enrolled to receive risdiplam orally once daily at a dose selected to achieve the targeted exposure range of close to 2000 ng*hr/mL.
Period: Overall Study
Arm/Group | 2 SMN2 Copies, Risdiplam | 3 SMN2 Copies, Risdiplam | >/=4 SMN2 Copies, Risdiplam
Started | 8 | 13 | 5
Primary Efficacy Population | 5 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 8 | 13 | 5
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Ongoing in Study | 5 | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 SMN2 Copies, Risdiplam | 3 SMN2 Copies, Risdiplam | >/=4 SMN2 Copies, Risdiplam | Total
Number analyzed (Participants) | 8 | 13 | 5 | 26
Age, Continuous [Mean (Standard Deviation); unit: days] | 22.8 (5.0) | 28.9 (7.5) | 31.2 (6.1) | 27.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 3 | 16
  Male | 4 | 4 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 5 | 12 | 5 | 22
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 11 | 3 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Two Copies of the Survival Motor Neuron (SMN) 2 Gene (Excluding the Known SMN2 Gene Modifier Mutation c.859G>C) and Baseline Compound Muscle Action Potential (CMAP) >=1.5 Millivolt (mV) Who Are Sitting Without Support
Description: The Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) Gross Motor Scale is a commonly used measure of infant and toddler development (0 to 42 months). The normed-scores derived from the BSID-III are used in clinical practice to detect infants with developmental delays, as well as to evaluate developmental progress and the impact of therapeutic interventions. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). Item 22, "sits without support for 5 seconds", is not considered achieved if the infant sits alone for less than 5 seconds before losing balance and falling over, or if the infant uses his or her arms to prop him- or herself up. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method. An exact binomial test was performed. If the lower limit of the two-sided 90% CI was above the 5% threshold, the primary objective of the study was considered achieved.
Time Frame: At Month 12
Population: Primary efficacy population included all infants in the intent-to-treat (ITT) population with two SMN2 copies (excluding the known SMN2 gene modifier mutation c.859G>C) and a baseline compound muscle action potential (CMAP) amplitude >/= 1.5 mV.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 2 SMN2 Copies, Risdiplam
Number analyzed (Participants) | 5
percentage of participants | 80.0 [34.26 to 98.98]
Statistical Analysis 1: Comparison: 2 SMN2 Copies, Risdiplam; Test type: Superiority; p < 0.0001, Exact Binomial Test; Performance Criterion = 5%

2. Secondary Outcome: Percentage of Participants Developing Clinically Manifested SMA
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

3. Secondary Outcome: Time to Permanent Ventilation and/or Death
Time Frame: Up to 7 years
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Participants Who Are Alive Without Permanent Ventilation
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Participants Alive
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants Who Achieve the Attainment Level of the Motor Milestones as Assessed in the Hammersmith Infant Neurological Examination-2 (HINE-2)
Description: HINE-2 assessment includes head control, sitting, voluntary grasp, ability to kick, rolling, crawling, standing, and walking
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Participants With Two Copies of the SMN2 Gene Sitting Without Support for 5 Seconds (Independent of the CMAP Value at Baseline).
Description: Assessed in Item 22 of the BSID-III Gross Motor Scale. The BSID-III is a commonly used measure of infant and toddler development (0 to 42 months). The normed-scores derived from the BSID-III are used in clinical practice to detect infants with developmental delays, as well as to evaluate developmental progress and the impact of therapeutic interventions. The gross motor scale consists of 72 items scored at 0 (unable to perform the activity) or 1 (criteria for item achieved). Item 22, "sits without support for 5 seconds", is not considered achieved if the infant sits alone for less than 5 seconds before losing balance and falling over, or if the infant uses his or her arms to prop him- or herself up. 90% CI for one sample binomial was computed using Clopper-Pearson (exact) method.
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population included all enrolled participants, regardless of whether they received risdiplam or not. Only participants with two copies of the SMN2 gene were included in this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 2 SMN2 Copies, Risdiplam
Number analyzed (Participants) | 8
percentage of participants | 87.5 [52.93 to 99.36]

8. Secondary Outcome: Percentage of Participants Sitting Without Support for 5 Seconds
Description: Assessed with BSID-III Gross Motor Scale
Time Frame: At Month 24
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Participants Sitting Without Support for 30 Seconds
Description: Assessed with BSID-III Gross Motor Scale
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

10. Secondary Outcome: Percentage of Participants Standing for at Least 3 Seconds
Description: Assessed with BSID-III Gross Motor Scale
Time Frame: At Month 24
Reporting Status: Not Posted

11. Secondary Outcome: Percentage of Participants Walking (Takes at Least 3 Steps)
Description: Assessed with BSID-III Gross Motor Scale
Time Frame: At Month 24
Reporting Status: Not Posted

12. Secondary Outcome: Percentage of Participants Demonstrating the Ability to Achieve a Scaled Score on BSID-III Gross Motor Subtests Within 1.5 Standard Deviations of Chronological Reference Standard
Description: Assessed through BSID-III Gross Motor Scale
Time Frame: At Month 24 and 42
Reporting Status: Not Posted

13. Secondary Outcome: Change From Baseline Score in the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Motor Function Scale at Month 12
Description: The CHOP-INTEND is a measure of motor function that was developed from the Test of Infant Motor Performance specifically for weak infants with neuromuscular disease. It consists of 16 items, where each item assesses a specific motor task (such as spontaneous movement of upper and lower extremity, hand grasping, rolling, head control, and others) graded on a scale of 0 to 4, where zero is no response and 4 is a complete response. A total score is calculated by summing the item scores (range 0 to 64) with lower scores indicating greater severity. A positive change from baseline indicates an improvement.
Time Frame: Baseline, Month 12
Population: ITT population included all enrolled participants, regardless of whether they received risdiplam or not.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | 2 SMN2 Copies, Risdiplam | 3 SMN2 Copies, Risdiplam | >/=4 SMN2 Copies, Risdiplam
Number analyzed (Participants) | 8 | 13 | 5
score on a scale
  Baseline | 46.50 [35.0 to 52.0] | 55.00 [44.0 to 62.0] | 50.00 [44.0 to 52.0]
  Change from Baseline at Month 12: number analyzed (Participants) | 8 | 13 | 4
  Change from Baseline at Month 12 | 9.50 [-6.0 to 20.0] | 8.00 [2.0 to 20.0] | 16.00 [8.0 to 19.0]

14. Secondary Outcome: Percentage of Participants Who Achieve a Score of 40 or Higher, 50 or Higher, and 60 or Higher in the CHOP INTEND Motor Function Scale at Month 12
Description: The CHOP-INTEND is a measure of motor function that was developed from the Test of Infant Motor Performance specifically for weak infants with neuromuscular disease. It consists of 16 items, where each item assesses a specific motor task (such as spontaneous movement of upper and lower extremity, hand grasping, rolling, head control, and others) graded on a scale of 0 to 4, where zero is no response and 4 is a complete response. A total score is calculated by summing the item scores (range 0 to 64) with lower scores indicating greater severity. Data are presented with a two-sided 90% Clopper-Pearson (exact) CI for the proportion.
Time Frame: At Month 12
Population: ITT population included all enrolled participants, regardless of whether they received risdiplam or not.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 2 SMN2 Copies, Risdiplam | 3 SMN2 Copies, Risdiplam | >/=4 SMN2 Copies, Risdiplam
Number analyzed (Participants) | 8 | 13 | 4
percentage of participants
  Score >=40 | 75.0 [40.03 to 95.36] | 100 [79.42 to 100.00] | 100 [47.29 to 100.00]
  Score >=50 | 75.0 [40.03 to 95.36] | 100 [79.42 to 100.00] | 100 [47.29 to 100.00]
  Score >=60 | 37.5 [11.11 to 71.08] | 100 [79.42 to 100.00] | 100 [47.29 to 100.00]

15. Secondary Outcome: Percentage of Participants Who Meet CHOP INTEND Stopping Criteria at Any Point
Time Frame: Up to Month 24
Reporting Status: Not Posted

16. Secondary Outcome: Change From Baseline in the Hammersmith Functional Motor Scale Expanded (HFMSE) Score
Time Frame: At Month 60
Reporting Status: Not Posted

17. Secondary Outcome: Number and Percentage of Participants Within 3rd Percentile of Normal Range for Weight-for-Age, Length/Height-for-Age and Weight-for-Length/Height
Description: Based on the WHO Child Growth Standards (WHO 2019)
Time Frame: At Month 12, 24, 36, 48 and 60
Reporting Status: Not Posted

18. Secondary Outcome: Number and Percentage of Participants Within 3rd Percentile of Normal Range for Head Circumference-for-age
Description: Based on the WHO Child Growth Standards (WHO 2019)
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

19. Secondary Outcome: Change From Baseline Percentiles for Weight-for-age, Length/Height-for-age, and weight-for- Length/Height
Time Frame: At Month 12, 24, 36, 48 and 60
Reporting Status: Not Posted

20. Secondary Outcome: Change From Baseline Percentiles for Head Circumference- For-age
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

21. Secondary Outcome: Change From Baseline in Chest Circumference
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

22. Secondary Outcome: Ratio Between Chest and Head Circumferences
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

23. Secondary Outcome: Percentage of Participants With the Ability to Swallow and to Feed Orally
Time Frame: At Month 12, 24, 36, 48 and 60
Reporting Status: Not Posted

24. Secondary Outcome: Change From Baseline in Compound Muscle Action Potential (CMAP) Amplitude
Description: Measured by CMAP
Time Frame: At Month 12 and 24
Reporting Status: Not Posted

25. Secondary Outcome: Measurement of Pharmacodynamic Marker Levels in Blood
Time Frame: Day 1, 56, 196, 364, 728 and at early withdrawal
Reporting Status: Not Posted

26. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Adverse event severity is determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5 (NCI CTCAE) v5
Time Frame: Up to 7 years
Reporting Status: Not Posted

27. Secondary Outcome: Ophthalmological Examination as Appropriate for Age
Time Frame: Up to 7 years
Reporting Status: Not Posted

28. Secondary Outcome: Plasma Concentration of Risdiplam and Its Metabolites to Characterize the PK Profile
Time Frame: Up to 7 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline up to the clinical cut off date (a minimum of 12 months and a maximum of 3.5 years)
Description: The safety population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not.
Arm/Group | 2 SMN2 Copies, Risdiplam | 3 SMN2 Copies, Risdiplam | >/=4 SMN2 Copies, Risdiplam
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/13 | 1/5
Other Adverse Events (participants affected / at risk) | 8/8 | 12/13 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 SMN2 Copies, Risdiplam (N=8) | 3 SMN2 Copies, Risdiplam (N=13) | >/=4 SMN2 Copies, Risdiplam (N=5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 SMN2 Copies, Risdiplam (N=8) | 3 SMN2 Copies, Risdiplam (N=13) | >/=4 SMN2 Copies, Risdiplam (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal pigmentation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Teething (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (7) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 4 (7) | 2 (5)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
COVID-19 (Infections and infestations) | 2 (2) | 7 (7) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (3)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (4) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (5)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Expired product administered (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Intercepted medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Underdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT03779334/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT03779334/SAP_001.pdf